CLINICAL TRIAL: NCT04453514
Title: Cultivating Calm During COVID-19: A Feasibility Study of Video-based Trauma-informed Yoga
Brief Title: Feasibility of a Brief Trauma-informed Yoga Intervention for Anxiety During the Coronavirus Disease (COVID-19) Pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Natural Medicine (Other)
Responsible Party: Principal Investigator, Deanne Tibbitts, PhD, Research Investigator, National University of Natural Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Tibbitts_TIYoga_COVID
Record Dates: First submitted 2020-06-30; First posted 2020-07-01 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Anxiety
Keywords: Yoga; Mind-Body Therapies; Complementary Therapies; Online
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trauma-informed yoga video recording (Experimental): Participants will complete a single trauma-informed yoga practice using a 45-minute guided video recording.
  Interventions: Behavioral: Trauma-informed yoga video recording

INTERVENTIONS:
Behavioral: Trauma-informed yoga video recording — Pre-recorded video of a 45-minute trauma-informed yoga practice. The yoga practice can be done standing or sitting in a chair. The yoga practice is comprised of slow, gentle movements combined with paying attention to the body and the breath. The practice uses invitational language and encourages participants to make choices and customize the movements according to their individual needs.

SUMMARY:
This study will help the investigators understand whether it is feasible and acceptable for people to practice trauma-informed yoga using a pre-recorded video. This study will also explore the immediate effects of trauma-informed yoga on anxiety, mindfulness, and body awareness. The results of this study will inform future research on remote delivery of trauma-informed yoga for supporting psychological wellbeing.

DETAILED DESCRIPTION:
Emerging data shows a high prevalence of anxiety during the first several months of the COVID-19 pandemic in the United States. Accordingly, there have been calls for supportive interventions for psychological health during the pandemic. Due to physical distancing requirements, supportive interventions for psychological health will be most accessible if they can be administered remotely. Trauma-informed yoga may support psychological health during the COVID-19 pandemic, but research on remote delivery of trauma-informed yoga is needed. The present study will evaluate the feasibility and acceptability of trauma-informed yoga delivered remotely. In this study, the investigators will create an online delivery platform within REDCap, a secure web application for research, that 1) hosts a 45-minute video of a trauma-informed yoga practice, and 2) collects data on participants' present moment experience of anxiety, mindfulness, and body awareness immediately before and after the yoga practice. Feasibility and acceptability data will allow the investigators to evaluate recruitment methods and refine the delivery method of trauma-informed yoga in a way that aligns with participant preferences. The investigators will also evaluate the short-term effects of trauma-informed yoga on state anxiety, state mindfulness, and body awareness. This study will allow the investigators to pilot the remote delivery of trauma-informed yoga during the ongoing, highly stressful COVID-19 pandemic and further develop trauma-informed yoga as a supportive intervention for psychological health.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Has an internet connection
* Willing to try a gentle yoga practice

Exclusion Criteria:

* Cannot read or understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2021-06-19 (Actual); Study Completion 2021-06-19 (Actual)

PRIMARY OUTCOMES:
Number of participants enrolled over 3 months | 3 months
  Total number of participants
Number of participants enrolled per week over 3 months | 3 months
  Count of participants enrolled each week
Proportion of participants who enroll in the study over 3 months | 3 months
  Proportion of participants who enroll out of the total who access the consent form
Proportion of participants who complete the study over 3 months | 3 months
  Proportion of participants that reach the final page of the study out of the total who provided informed consent
Proportion of missing data over 3 months | 3 months
  Proportion of participants who filled out less than 70% of the items per questionnaire; mean proportion of items skipped per questionnaire
Proportion of participants who complete the 45-minute video over 3 months | 3 months
  Proportion of participants who self-report watching the video in its entirety and for whom time stamps show that the time elapsed on the page where the video is embedded is greater than or equal to 80% of the length of the video

SECONDARY OUTCOMES:
Mean change in state anxiety from immediately before to immediately after yoga using the State Trait Anxiety Scale - 6 item short form | immediately before/after
  The State Trait Anxiety Inventory (STAI) - Y6 is a 6-item, validated self-report questionnaire that assesses state anxiety when used with instructions that specify: "indicate how you feel right now, in this moment." Responses to each item are provided on a 4 point Likert Scale ('Not at all' to 'Very much'). The instrument is scored as the mean of 6 items, multiplied by 20 to use the interpretation guide for the full STAI scale.
Mean change in state mindfulness from immediately before to immediately after yoga using the State Mindfulness Scale (State Mindfulness of Mind subscale) | immediately before/after
  The State Mindfulness Scale is a 21-item, validated self-report questionnaire that assesses state mindfulness. The State Mindfulness Scale is comprised of two subscales, State Mindfulness of Mind and State Mindfulness of Body. Responses to each item are provided on a 5 point Likert Scale ('Not at all' to 'Very much'). The instrument is scored as the sum of scores from each subscale. For this outcome, the State Mindfulness of Mind subscale will be used.
Mean change in body awareness from immediately before to immediately after yoga using the State Mindfulness Scale (State Mindfulness of Body subscale) | immediately before/after
  The State Mindfulness Scale is a 21-item, validated self-report questionnaire that assesses state mindfulness. The State Mindfulness Scale is comprised of two subscales, State Mindfulness of Mind and State Mindfulness of Body. Responses to each item are provided on a 5 point Likert Scale ('Not at all' to 'Very much'). The instrument is scored as the sum of scores from each subscale. For this outcome, the State Mindfulness of Body subscale will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Deanne Tibbitts, PhD, Principal Investigator — National University of Natural Medicine
Locations (1):
- National University of Natural Medicine, Portland, Oregon, United States